CLINICAL TRIAL: NCT00193414
Title: Phase II Study of First-Line Therapy With Pemetrexed and Gemcitabine in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Pemetrexed and Gemcitabine in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 91; H3E-US-X011
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2012-11-13 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Chemotherapy-naïve patients with unresectable stage III/IV NSCLC received pemetrexed 500 mg/m2 IV and gemcitabine 1500 mg/m2 IV every 2 weeks for 8-12 cycles with restaging every 4 cycles. Patients also received supplemental folate/B12 therapy.
  Interventions: Drug: Pemetrexed; Drug: Gemcitabine

INTERVENTIONS:
Drug: Pemetrexed — 500mg/m2 IV over 10 min, Day 1, prior to gemcitabine
  Other Names: Alimta
Drug: Gemcitabine — 1500mg/m2, 30min IV
  Other Names: Gemzar

SUMMARY:
This study is designed to study the role of an active and well-tolerated non-platinum agent, gemcitabine, in a combination regimen with pemetrexed in the first-line treatment of advanced NSCLC. This study will serve to define the role of next generation agents in a new combination regimen in the treatment of advanced NSCLC. This combination regimen may ultimately be important in further expanding treatment options for patients while improving survival, quality of life, and symptom control compared with platinum-based combination regimens - and with acceptable toxicity.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be receive:

* Pemetrexed + Gemcitabine

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Histologically confirmed non-small cell bronchogenic carcinoma
* Newly diagnosed or recurrent unresectable stage III or stage IV disease
* No mixed tumors with small cell anaplastic elements
* Measurable disease
* Must not have received any prior antineoplastic chemotherapy for lung cancer
* Age > 18 years
* Able to perform activities of daily living with little or no assistance
* Adequate bone marrow, liver and kidney
* Understand the nature of this study and give written informed consent.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Female patients who are pregnant or are lactating
* History of serious cardiovascular disease within the previous six months
* Serious active infection at the time of treatment
* Other serious underlying medical condition

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-05; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, Nashville, Tennessee, United States

REFERENCES:
- [Result] Spigel DR, Hainsworth JD, Barton JH, Patton JF, Zubkus JD, Simons L, Griner P, Burris HA 3rd, Greco FA. Phase II study of biweekly pemetrexed and gemcitabine in patients with previously untreated advanced non-small cell lung cancer. J Thorac Oncol. 2010 Jun;5(6):841-5. doi: 10.1097/JTO.0b013e3181d737e3. PMID 20421819
- See also: Published article in the Journal of Thoracic Oncology — http://journals.lww.com/jto/pages/articleviewer.aspx?year=2010&issue=06000&article=00015&type=abstract

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 72
Completed | 14
Not Completed | 58

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 47
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate is the percentage of patients with complete response or partial response per RECIST v.1 Criteria. Complete response (CR) = Disappearance of all target lesions, disappearance of all nontarget lesions for at least 4 weeks. Partial Response (PR) = At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameters.
Time Frame: 18 months
Population: All patients were assessed for response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Intervention
Number analyzed (Participants) | 72
Percentage of participants | 26 [17 to 38]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the interval between the start date of treatment and the date of occurrence of progressive disease or death from any cause.
Time Frame: 18 months
Population: All patients were assessed for PFS.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intervention
Number analyzed (Participants) | 72
Months | 6.2 [4.1 to 8.1]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was measured from the date of study entry until the date of death.
Time Frame: 18 months
Population: All patients were assessed for OS.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intervention
Number analyzed (Participants) | 72
Months | 8.5 [6.7 to 11.5]

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 39/72
Other Adverse Events (participants affected / at risk) | 72/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=72)
Altered Mental Status (Nervous system disorders) | 1
Cardiac General - Other (Congestive Heart Failure) (Cardiac disorders) | 1
Cardiac ischemia/infarction (Cardiac disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Death not associated with CTCAE term - Disease Progression NOS (General disorders) | 17
Pancreatic endocrine: glucose intolerance (Endocrine disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (General disorders) | 1
Febrile Neutropenia (Infections and infestations) | 3
Fever (General disorders) | 1
Fracture (Limb) (Musculoskeletal and connective tissue disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 2
Hemorrhage, GI (Blood and lymphatic system disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypoxemia (General disorders) | 3
Infection - Other (Cellulitis) (Infections and infestations) | 3
Infection - Other (Pneumonia) (Infections and infestations) | 8
Leukocytes (Blood and lymphatic system disorders) | 1
Neurology - Other (Spinal Cord Compression) (Nervous system disorders) | 1
Pain - Gastrointestinal (Gastrointestinal disorders) | 1
Pain - NOS (General disorders) | 1
Pancytopenia (NOS) (Blood and lymphatic system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory - Other (Post obstructive lung process) (Respiratory, thoracic and mediastinal disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Seizure (Nervous system disorders) | 1
Supraventricular and nodal arrhythmia - Atrial Arrhythmia (NOS) (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia - Atrial Fibrillation (Cardiac disorders) | 4
Supraventricular and nodal arrhythmia - Atrial Flutter (Cardiac disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 6
Supraventricular and nodal arrhythmia - Supraventricular tachycardia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=72)
Alopecia (Skin and subcutaneous tissue disorders) | 16
Anorexia (Gastrointestinal disorders) | 31
Pain - Joints (Musculoskeletal and connective tissue disorders) | 8
Fatigue (General disorders) | 72
Cardiac Toxicity (Cardiac disorders) | 7
Diarrhea (Gastrointestinal disorders) | 14
Edema (Blood and lymphatic system disorders) | 33
Febrile Neutropenia (Infections and infestations) | 8
Fever (General disorders) | 20
Hypotension (Cardiac disorders) | 5
Infection (NOS) (Infections and infestations) | 33
Mucositis (Gastrointestinal disorders) | 16
Pain - muscles (Musculoskeletal and connective tissue disorders) | 8
Nausea (Gastrointestinal disorders) | 38
Pain - NOS (General disorders) | 32
Peripheral Neuropathy NOS (Nervous system disorders) | 5
Pulmonary symptoms (Cardiac disorders) | 16
Skin Toxicity (Skin and subcutaneous tissue disorders) | 32
Vomiting (Gastrointestinal disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at the site.